CLINICAL TRIAL: NCT03963986
Title: Impacts of Remote Digital Support on Adapted Physical Activity for Patients in Pre-bariatric Surgery Care Pathways
Brief Title: Impacts of Remote Digital Support on Physical Activity for Patients in Bariatric Surgery
Acronym: STIMUL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STIMUL
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Bariatric Surgery
Keywords: Regular physical activity

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to the STANDARD group for which management will be standard or to the STIMUL group with digital coaching program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STIMUL group (Active Comparator): The STIMUL Group participants in the Adaptive Physical Activity Focus (APA) program receive access to an online digital Platform, as well as a starter kit consisting of a connected pedometer measuring several physical activity indicators including the number of steps, number of so-called active minutes, sleep time, and distance travelled; a tape measure and a starter guide. They then conduct a remote assessment and motivational interview by videoconference or telephone, followed by 15-20 minute support interviews (month 1, month 3, month 6). Between these interviews, during months 1, 2, and 3, participants exchange weekly written messages with an educator on their platform. A planner of their physical activity objectives is provided.
  Interventions: Device: STIMUL group
- STANDARD group (No Intervention): The STANDARD group participants dont receive an access to an online digital platform but they receive an adapted advice sheet.

INTERVENTIONS:
Device: STIMUL group — The STIMUL Group participants in the Adaptive Physical Activity Focus (APA) program receive access to an online digital Platform, as well as a starter kit consisting of a connected pedometer measuring several physical activity indicators including the number of steps, number of so-called active minutes, sleep time, and distance travelled; a tape measure and a starter guide. They then conduct a remote assessment and motivational interview by videoconference or telephone, followed by 15-20 minute support interviews (month 1, month 3, month 6). Between these interviews, during months 1, 2, and 3, participants exchange weekly written messages with an educator on their platform. A planner of their physical activity objectives is provided.
  Arms: STIMUL group

SUMMARY:
Compare the level of PA (physical activity) in groups with and without STIMUL device at 4 months

DETAILED DESCRIPTION:
Regular physical activity (PA) is a key element in the success of bariatric surgery and the prevention of complications associated with frequent co-morbidities. However, the levels of PA observed in patients who will benefit from bariatric surgery are generally low, and many patients do not comply with the recommendations of their course in terms of PA. It is envisaged that coaching interventions and adapted programs can improve the level of PA. The objective of this pilot study is to evaluate the effectiveness and adherence to digital tools on the level of PA in preparation for bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 30 to 50 years.
* Candidate for bariatric surgery within 4 to 6 months of inclusion: BMI >40 kg/m² or BMI 35-40 kg/m² with obesity-related comorbidity
* Ability to follow the STIMUL education program focused on adapted physical activity
* Has and knows how to use a computer connected to the Internet or mobile phone
* Ability to understand, read and write French

Exclusion Criteria:

* • Contra-indication to the practice of sport

  * refusal to participate in the study
  * refusal to participate in the study

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Ricci-Gagnon score (9-45) | month 4
  This score describe the physical profile : inactive, active, very active, at month 4 It is calculated by adding the number of points (1 to 5) corresponding to the box checked for each question.
  Less than 18=inactive Between 18 and 35=active More than 35=Active

SECONDARY OUTCOMES:
Ricci-Gagnon score (9-45) | 10 and 16 months
  This score describe the physical profile : inactive, active, very active, at month 10 et 16 It is calculated by adding the number of points (1 to 5) corresponding to the box checked for each question.
  Less than 18=inactive Between 18 and 35=active More than 35=Active
International Physical Activity Questionnaire (IPAQ) | 4, 10 and 16 months
  physical activity score
  1. - LowNo activity is reported ORAn activity is reported but does not reach levels 2 or 3.
  2. -ModerateCorresponds to one of the following 3 criteria:3 days or more of intense activity for at least 20 min per day OR5 days or more of moderate intensity activity and/or walking for at least 30 min per day OR5 days or more of combined walking, moderate or high intensity activity, reaching at least 600 MET-minutes/week
  3. -HighCorresponds to one of the following 2 criteria:Intense activity at least 3 days per week and at least 1500 MET-minutes/week OR 7 or more days of combined walking, moderate or high intensity activity, reaching at least 3000 MET-minutes/week.
Body masse Index (BMI) (kg/m²) | 4, 10 and 16 months
  Comparison of BMI in the 2 groups at 4, 10, and 16 months BMI < 18.5 kg/m²: underweight 18.5 < BMI < 24.9: normal weight 25 < BMI < 29.9: overweight BMI > 30: obesity
Waist circumference (cm) | 4, 10 and 16 months
  Comparison of waist circumference in the 2 groups at 4, 10, and 16 months
Hip circumference (cm) | 4, 10 and 16 months
  Comparison of waist circumference in the 2 groups at 4, 10, and 16 months
Lipid balance (g/l) | 4, 10 and 16 months
  Evolution of the lipid balance in the 2 groups
Blood pressure (mmHg) | 4, 10 and 16 months
  Evolution of blood pressure in the 2 groups
Quality of Life, Obesity and Dietetics Scale(EQVOD) | 4, 10 and 16 months
  Evolution of the quality of life (EQVOD)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No